CLINICAL TRIAL: NCT00126334
Title: Conservative Versus Liberal Red Cell Transfusion in Myocardial Infarction Trial: The CRIT Pilot
Acronym: CRIT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Dr. Neil Weissman, Medstar Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2003-003
Record Dates: First submitted 2005-08-02; First posted 2005-08-03 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-07

CONDITIONS: Myocardial Infarction; Anemia
Keywords: Myocardial Infarction; Anemia; Erythrocyte Transfusion
MeSH Terms: conditions — Myocardial Infarction; Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Liberal transfusion threshold
  Interventions: Procedure: Packed Red Blood Cell Transfusion
- 2 (Experimental): Conservative transfusion threshold
  Interventions: Procedure: Packed Red Blood Cell Transfusion

INTERVENTIONS:
Procedure: Packed Red Blood Cell Transfusion — transfusion of 1 unit of PRBCs

SUMMARY:
The purpose of this trial is to determine whether a conservative or a liberal blood transfusion strategy is better for patients with a heart attack and a low blood count.

DETAILED DESCRIPTION:
The current standard of care for patients with heart attacks is to transfuse red blood cells when the hematocrit (red blood cell count) drops below 30 percent. However, there is little scientific basis for this current standard, and recent research has demonstrated that it is safe to allow the hematocrit (red blood cell count) to drop significantly lower in severely ill medical patients and in patients with heart disease undergoing major surgery. The investigators therefore propose this pilot trial to begin to determine whether or not it is safe to apply a more conservative blood transfusion strategy to patients with heart attacks.

In this study, patients who are within 72 hours of the onset of a heart attack and who are anemic (have a low red blood cell count) will be randomly assigned to one of two transfusion strategies while they are in the hospital: a liberal strategy of transfusing blood when the hematocrit falls below 30 percent (the current standard) or a conservative strategy of transfusing blood only when the hematocrit falls below 24 percent. It will then be determined which group fares better over the next 30 days.

The plan is to enroll 92 patients in this pilot trial in order to allow the researchers to plan for a much larger, definitive trial of this important question. It is anticipated that the conservative transfusion strategy will be similar to the standard (liberal) strategy in terms of patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

All of the following must be present:

* Acute myocardial infarction with presentation within 72 hours of randomization (acute myocardial infarction is defined as ischemic-type chest discomfort lasting at least 30 minutes associated with creatinine kinase MB (CKMB) or troponin >upper limit of normal [ULN])
* Admission to CCU
* Hematocrit .30 or less
* Written, informed consent

Exclusion Criteria:

* Inability or unwillingness to receive red cell transfusions
* Active bleeding (overt blood loss accompanied by a decrease in hematocrit of at least 5% in the preceding 12 hours)
* Receipt of red cell transfusion within 7 days of randomization
* Prior severe transfusion reaction
* Pregnancy
* Imminent death
* Decision to provide limited care
* Age <21
* Participation in another clinical trial in which blood transfusion is a requirement or a component of a primary or secondary endpoint
* Previous participation in the CRIT Pilot

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2003-04; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
In-hospital death | In-hospital
Recurrent myocardial infarction (MI) | In-hospital
New or worsening heart failure | In-hospital

SECONDARY OUTCOMES:
Critical Care Unit (CCU) length of stay | In-hospital
Length of hospitalization | In-hospital
Death or recurrent MI at hospital discharge and 30 days | 30 days
Death or recurrent MI or new or worsening congestive heart failure (CHF) at 30 days | 30 days
Death at 30 days | 30 days
In-hospital recurrent ischemia | In-hospital
In-hospital death or recurrent MI or new or worsening CHF or recurrent ischemia | In-hospital
Acute renal insufficiency (increase in serum creatinine of ≥ 0.5mg/dL) | In-hospitall
Number of transfusions received per patient | In-hospital
Proportion of patients receiving at least one transfusion | In-hospital
Mean daily hematocrit | In-hospital
Transfusion-related reactions | In-hospital

CONTACTS AND LOCATIONS:
Overall Officials: Howard A Cooper, M.D., Principal Investigator — Medstar Health Research Institute
Locations (3):
- United States (3):
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Washington VA Medical Center, Washington D.C., District of Columbia
  - Durham VA Medical Center, Durham, North Carolina

REFERENCES:
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Fergusson DA, Pagano MB, Roubinian NH, Turgeon AF, Valentine S, Trivella M, Doree C, Hebert PC. Transfusion thresholds and other strategies for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2025 Oct 20;10(10):CD002042. doi: 10.1002/14651858.CD002042.pub6. PMID 41114449
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Trivella M, Roubinian N, Fergusson DA, Triulzi D, Doree C, Hebert PC. Transfusion thresholds for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2021 Dec 21;12(12):CD002042. doi: 10.1002/14651858.CD002042.pub5. PMID 34932836